CLINICAL TRIAL: NCT06266273
Title: Investigating the Development, Validity, and Reliability of the Avoidance of Sports Activities Photo Scale
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Turgut, Associate Professor Elif TURGUT, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SBA 23/442
Record Dates: First submitted 2024-02-01; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Questionnaire; Athletes; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Overhead athletes with shoulder pain (Other): * Male and female athletes aged between 18-35,
  * Engaged professionally in sports involving overhead activities for at least 3 years (volleyball, basketball, swimming, badminton, water polo, tennis, American football, handball, etc.),
  * Actively participating in competitions for at least 1 year,
  * Experiencing current traumatic or non-traumatic pain, or having a history of shoulder pain, or having chronic shoulder pain
  * Native Turkish speakers.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
"Investigating the Development, Validity, and Reliability of the Avoidance of Sports Activities Photo Scale" is crucial in determining the specific functional status of the shoulder joint, especially for overhead athletes experiencing shoulder pain, to identify which sporting activities restrict them the most and to fill the gap in the literature. Additionally, visually indicating activities through photographs will provide visual feedback, making it easier to assess functional status. Our study aims to develop a specific functional survey for the shoulder joint in overhead athletes, examine the validity and reliability of this scale, and contribute to the literature.

DETAILED DESCRIPTION:
Developing a valid and reliable visual assessment scale specifically targeting shoulder pain in overhead athletes with shoulder pain, aiming to evaluate shoulder pain in a specific and functional manner, and investigating its psychometric properties.The research will be conducted at Hacettepe University Faculty of Physical Therapy and Rehabilitation, Athlete Health Unit. The research will be conducted according to the Consensus-Based Standards for the Selection of Health Measurement Instruments (COSMIN) guidelines. COSMIN guidelines recommend a minimum of 100 participants for reliability, measurement error, and validity assessments. Therefore, the study plans to include at least 100 individuals who apply to the Athlete Health Unit at Hacettepe University Faculty of Physical Therapy and Rehabilitation. The data collection for this planned study will be solely through surveys. The design of the study is a cross-sectional study aimed at developing and assessing the validity and reliability of the "Avoidance of Sports Activities Photo Scale." Surveys specific to the research will be implemented in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female athletes aged between 18-35,
* Engaged professionally in sports involving overhead activities for at least 3 years (volleyball, basketball, swimming, badminton, water polo, tennis, American football, handball, etc.),
* Actively participating in competitions for at least 1 year,
* Experiencing current traumatic or non-traumatic pain, or having a history of shoulder pain, or having chronic shoulder pain,
* Native Turkish speakers.

Exclusion Criteria:

* Neurological and/or rheumatological disease,
* Active local or systemic infection,
* History of cancer,
* Severe visual impairment.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Investigating the Development, Validity, and Reliability of The Sports Activity Avoidance Photo Scale | 10-15 minutes for each participant
  Investigation, validity and reliability of the Sports Activity Avoidance Photo Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Elif Turgut, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No